CLINICAL TRIAL: NCT07176273
Title: Changing the Treatment Course: Clinical Trial of Sequenced Interventions to Optimize Treatment for Veterans With PTSD
Brief Title: Adaptive Decision-making And Personalized Treatment for PTSD (ADAPT-PTSD)
Acronym: ADAPT-PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stefanie LoSavio, Assistant Professor of Psychiatry & Behavioral Sciences, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001551; HT9425-24-1-1026 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Posttraumatic Stress Disorder; PTSD
Keywords: Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled effectiveness trial utilizing a Hybrid Experimental Design (HED) comprised of a Sequential Multiple Assignment Randomized Trial (SMART) and Micro-Randomized Trial (MRT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Early CPT Non-Responders Switch (Group A) (Active Comparator): Early NON-RESPONDERS to CPT will SWITCH to PE
  Interventions: Behavioral: Digital Interventions; Behavioral: Cognitive Processing Therapy (CPT); Behavioral: Prolonged Exposure (PE)
- Early CPT Non-Responders Modular (Group B) (Active Comparator): Early NON-RESPONDERS to CPT will transition to MODULAR CPT
  Interventions: Behavioral: Modular Cognitive Processing Therapy; Behavioral: Digital Interventions; Behavioral: Cognitive Processing Therapy (CPT)
- Early CPT Responders Continue (Group C) (Active Comparator): Early RESPONDERS to CPT will CONTINUE in their CPT treatment
  Interventions: Behavioral: Digital Interventions; Behavioral: Cognitive Processing Therapy (CPT)
- Early CPT Responders Step Down (Group D) (Active Comparator): Early RESPONDERS to CPT will STEP DOWN to self-managed CPT
  Interventions: Behavioral: Step Down Treatment; Behavioral: Digital Interventions; Behavioral: Cognitive Processing Therapy (CPT)
- Early PE Non-Responsers Switch (Group E) (Active Comparator): Early NON-RESPONDERS to PE will SWITCH to CPT
  Interventions: Behavioral: Digital Interventions; Behavioral: Cognitive Processing Therapy (CPT); Behavioral: Prolonged Exposure (PE)
- Early PE Non-Responders Modular (Group F) (Active Comparator): Early NON-RESPONDERS to PE will transition to MODULAR PE
  Interventions: Behavioral: Modular Prolonged Exposure Therapy; Behavioral: Digital Interventions; Behavioral: Prolonged Exposure (PE)
- Early PE Responders Continue (Group G) (Active Comparator): Early RESPONDERS will CONTINUE in their PE treatment
  Interventions: Behavioral: Digital Interventions; Behavioral: Prolonged Exposure (PE)
- Early PE Responders Step Down (Group H) (Active Comparator): Early RESPONDERS to PE will STEP DOWN to self-managed PE
  Interventions: Behavioral: Step Down Treatment; Behavioral: Digital Interventions; Behavioral: Prolonged Exposure (PE)

INTERVENTIONS:
Behavioral: Modular Cognitive Processing Therapy — CPT is a first-line treatment for PTSD that includes the following core elements: (a) identification of "stuck points" in thinking that interfere with recovery and (b) using Socratic questioning and a series of Contains the same core elements of CPT, but content is repackaged into modules instead of sessions so that clinicians can select and dose treatment elements according to patient need. Modular CPT contains the same core elements of CPT, but content is repackaged into modules instead of sessions so that clinicians can select and dose treatment elements according to patient need.
  Other Names: Modular CPT
  Arms: Early CPT Non-Responders Modular (Group B)
Behavioral: Modular Prolonged Exposure Therapy — PE is a first-line treatment for PTSD that includes the following core elements: (a) in vivo exposure and (b) imaginal exposure to the trauma memory. Modular PE is comprised of the same elements of standard PE, but clinicians select and dose modules (i.e., imaginal exposure, in vivo exposure) based on individual patient need.
  Other Names: Modular PE
  Arms: Early PE Non-Responders Modular (Group F)
Behavioral: Step Down Treatment — Self-managed treatment will involve receiving a self-help version of the remaining treatment materials and ongoing use of the intervention companion app (CPT Coach or PE Coach).
  Other Names: Step Down
  Arms: Early CPT Responders Step Down (Group D); Early PE Responders Step Down (Group H)
Behavioral: Digital Interventions — The prompt will be a text message delivered through VA-approved technology (e.g., PETALS).
  Other Names: Daily Digital Prompts
Behavioral: Cognitive Processing Therapy (CPT) — CPT is a first-line treatment for PTSD that includes the following core elements: (a) identification of "stuck points" in thinking that interfere with recovery and (b) using Socratic questioning and a series of progressive worksheets to examine stuck points, develop balanced beliefs, and facilitate the experience of natural emotions.
  Other Names: CPT
  Arms: Early CPT Non-Responders Modular (Group B); Early CPT Non-Responders Switch (Group A); Early CPT Responders Continue (Group C); Early CPT Responders Step Down (Group D); Early PE Non-Responsers Switch (Group E)
Behavioral: Prolonged Exposure (PE) — PE is a first-line treatment for PTSD that includes the following core elements: (a) in vivo exposure and (b) imaginal exposure to the trauma memory. In imaginal exposure, participants repeatedly, systematically approach their trauma memory and related thoughts and feelings. In in vivo exposure, participants repeatedly, systematically approach objectively safe people, places, objects, and situations that they avoid because these stimuli remind them of their trauma.
  Other Names: PE
  Arms: Early CPT Non-Responders Switch (Group A); Early PE Non-Responders Modular (Group F); Early PE Non-Responsers Switch (Group E); Early PE Responders Continue (Group G); Early PE Responders Step Down (Group H)

SUMMARY:
By doing this research project, the investigators hope to learn which strategies work best to help veterans who are not benefiting from their first PTSD treatment or not completing between-session homework assignments regularly that might improve treatment response. The investigators also want to learn how best to match the right type and amount of treatment to each individual veteran. By conducting this research project, they hope to:

* See if trying a different treatment strategy for veterans not responding to their first PTSD treatment would be more helpful
* See if sending text message prompts between sessions encourages more completion of between-session homework

DETAILED DESCRIPTION:
This study is designed to assist the investigators in answering the clinical question of how to address non-response to first line PTSD treatments. Utilizing an innovative Hybrid Experimental Design (HED), the proposed study involves multiple, sequential randomizations to both therapist-delivered and digital interventions operating on short and long timescales to determine the optimal combination and sequencing of evidence-based interventions to maximize response. This will result in actionable data and, consistent with a personalized medicine approach, an implementable, adaptive treatment regimen that optimizes clinical resource allocation. By recruiting and providing treatment in routine care settings serving veterans with PTSD, the study design maximizes generalizability, relevance to the VA mission, and implementation potential.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans eligible for PE and CPT at the participating PTSD treatment-providing clinic who are
2. At least 18 years or older
3. Score ≥ 31 on the PCL-5 secondary to a Criterion A traumatic event
4. Own a mobile device that can be used for the therapy companion mobile app (Prolonged Exposure (PE) coach or Cognitive Processing Therapy (CPT) coach).

Exclusion Criteria:

1. Acute suicide risk requiring clinical intervention
2. Need for detoxification
3. Unmanaged psychosis or bipolar disorder
4. Severe cognitive impairment that makes it unlikely that participants can adhere to the study regimen (as evidenced by confusion, inability to track discussion or answer questions, or other clear and significant indicators of cognitive impairment)
5. Current or past 12-month engagement in PE or CPT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2028-05-22 (Estimated); Study Completion 2028-08-14 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist (PCL-5) | 10 weeks, 20 weeks and 9 months
  The PCL-5 is a psychometrically valid measure and commonly used assessment of PTSD symptoms. A total score is calculated by adding up the ratings for each of the 20 items, which range from 0 to 4 (0=Not at all, 4=Extremely). Higher scores reflect more severe symptoms. A score below 31 generally suggests a sub-clinical range, while scores of 31 or above fall within the clinical range, indicating probable PTSD.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 10-weeks, 20-weeks, 9-months
  The PHQ-9 score indicates the severity of depressive symptoms. There are 9 items with scores ranging from 0-3 for each. Total scores range from 0 to 27, with higher scores indicating more severe symptoms. A score of 5-9 is considered mild, 10-14 is moderate, 15-19 is moderately severe, and 20-27 is severe. The PHQ-9 score is not a diagnosis, but rather a screening tool to assess depression severity and guide treatment decisions.
Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline, 10-weeks, 20-weeks, 9-months
  The C-SSRS is a standardized measure used to assess suicide risk, primarily through the presence and severity of suicidal ideation and behavior. The screener version of the C-SSRS consists of 2-6 "Yes" or "No" questions. Responses to questions 1 and 2 determine if questions 3, 4, and 5 are asked. A 'Yes' answer to question 2 prompts questions 3, 4, 5, and 6. A 'No' answer to question 2 directs the responder to question 6. Affirmative ("Yes") responses are summed, with each 'Yes' counting as 1 point. This summation provides a score on a scale of 0-6 indicating suicide risk level.
  0 = No risk reported (all "No" responses).
  1 - 2 = Low risk. 3 - 6 = Moderate to high risk. A "Yes" response to question 3 or 6a indicates moderate risk (potential plan or lifetime engagement in preparatory behavior). A "Yes" response to question 4, 5, or 6b indicates high risk (active plan, possible intent, or recent preparatory behaviors).
Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) | Baseline, 20-weeks, 9-months
  The Q-LES-Q-SF contains 16 questions scored on a 5-point Likert scale with values from 1 ("Very Poor") to 5 ("Very Good"). A total score is calculated by summing the first 14 item responses and ranges from 14 to 70; higher scores are associated with greater life satisfaction and enjoyment. The total score is expressed as a percentage based on the maximum total score of the items completed (1-100). The normal range that represents community sample scores is 70-100, and thus scores below 70 are clinically significant. Note, the last two items (items 15 and 16) ask about medication and overall contentment and are stand-alone items; they are not included in the total score.
Brief Inventory of Psychosocial Functioning (B-IPF) | Baseline, 10-weeks, 20-weeks, 9-months
  The B-IPF is a 7-item self-report instrument that evaluates PTSD-related psychosocial functional impairment within the last 30 days across seven functional domains (romantic relationships, family relationships, work, friendships and socializing, parenting, education, and self-care). Items on the B-IPF are scored on a Likert scale from 0 (never) to 6 (always). The B-IPF was designed so that respondents complete only temporally relevant items that reflect a domain that they have participated in over the past 30 days (e.g., participants who were not enrolled in school within the past 30 days are instructed to skip the education item). The BIPF is scored by summing the scored items to create a total score, dividing the total score by the maximum possible score based on the number of items scored, and multiplying by 100. Thus, the B-IPF represents an overall index of functioning, with higher scores indicating greater functional impairment

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie LoSavio, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Rebecca Sripada, PhD, Principal Investigator — VA Ann Arbor-506
Locations (4):
- United States (4):
  - Augusta VA, Augusta, Georgia
  - Ann Arbor VA, Ann Arbor, Michigan
  - Battle Creek VA, Battle Creek, Michigan
  - Salt Lake City VA, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No